CLINICAL TRIAL: NCT00973622
Title: Changing Thought and Action in Tobacco Dependence With Transcranial Magnetic Stimulation
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 110881
Record Dates: First submitted 2009-08-26; First posted 2009-09-09 (Estimated); Results first posted 2013-09-24 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-07

CONDITIONS: Tobacco Dependence
Keywords: Tobacco cessation; Tobacco dependence; Transcranial Magnetic Stimulation; Nicotine Dependence; Delayed Discounting
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smokers (Experimental): Healthy adult smokers aged 19-55 who are not currently interested in quitting smoking.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS) 10 Hertz (Hz); Device: repetitive transcranial magnetic stimulation (rTMS) 20Hz; Device: SHAM repetitive transcranial magnetic stimulation (rTMS)
- Non-smokers (Experimental): Healthy adult non-smokers aged 19-55
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS) 10 Hertz (Hz); Device: repetitive transcranial magnetic stimulation (rTMS) 20Hz; Device: SHAM repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) 10 Hertz (Hz) — All participants will receive 90 10-pulse trains of 1 sec duration with an interval of 20 seconds. Smokers will receive the treatment twice, once in a nicotine-satiated condition, and once in a nicotine-withdrawal condition.
  Other Names: "TMS" or Transcranial Magnetic Stimulation
Device: repetitive transcranial magnetic stimulation (rTMS) 20Hz — All participants will receive 45 20-pulse trains of 1 second duration with an interval of 20 seconds. Smokers will receive the treatment twice, once in a nicotine-satiated condition, and once in a nicotine-withdrawal condition.
  Other Names: "TMS" or Transcranial Magnetic Stimulation
Device: SHAM repetitive transcranial magnetic stimulation (rTMS) — The look and sound of active rTMS is reproduced with the same coil used in the active conditions. The magnetic field in the sham coil is markedly attenuated at only 5% of stimulator output. The feel of active stimulation will be reproduced by delivering monophasic current pulses to the left, frontalis muscle with a Isolated Stimulator and two carbon rubber electrodes. Smokers will receive Sham rTMS in both the nicotine-satiated and nicotine-withdrawal conditions.
  Other Names: "TMS" or Transcranial Magnetic Stimulation

SUMMARY:
This study will examine the effects of high frequency, repetitive Transcranial Magnetic Stimulation (rTMS) on decision-making and smoking behavior.

DETAILED DESCRIPTION:
Tobacco use is the greatest cause of preventable death in the US and cigarette smokers exhibit substantial relapse following treatment. Understanding the brain mechanisms involved in tobacco dependence is an important step toward reducing the high rate of relapse associated with current behavioral and pharmacological treatments for smoking cessation. This study seeks to examine the effects of high frequency, repetitive Transcranial Magnetic Stimulation (rTMS) on decision-making and smoking behavior. A concept central to this study is that "quitting" tobacco necessitates making conscious choices not to smoke (to delay gratification) and these choices are influenced by the balance of activity between the frontal-parietal systems that process the value of rewards and limbic systems that are involved with immediate gratification. We aim to: 1) determine how two different levels of cortical excitation (10 Hz and 20Hz), induced by different rTMS frequencies, influence reward and risk-taking choices and cigarette consumption. Additionally, we aim to 2) determine how limbic activation due to acute nicotine withdrawal and/or satiation modifies the effects in aim 1. Twenty non-smoking and 20 smoking participants will receive two levels of high frequency rTMS and comparable sham stimulation (using electrical scalp stimulation) delivered over the left prefrontal cortex. Smokers will also crossover between nicotine satiation and acute withdrawal conditions to determine how rTMS interacts with limbic activation associated with nicotine use and withdrawal. In addition, changes in preattentional (brainstem-thalamus processing as measured using the P50 midlatency auditory evoked potential) and attentional (thalamocortical processing as measured using the Psychomotor Vigilance Task; PVT) will be assessed before and after treatment to quantitatively determine changes in preattentional/arousal and attentional function.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-55
* Must speak English
* Must be right handed
* Must pass the Transcranial Magnetic Stimulation Adult Safety and Screening Questionnaire (TAAS)
* Smoking participants must be highly dependent with a score of 6 or greater on the Fagerstrom Test for Nicotine Dependence

Exclusion Criteria:

* Positive test for drugs of abuse
* Positive pregnancy test
* A personal or family history of epilepsy
* A history of anticonvulsant medication use
* A personal history of head injury
* A history of aneurysm, stroke, or previous cranial neurosurgery
* A diagnosis of bipolar disorder
* A neurological or psychiatric disorder for which hospitalization was required
* Tinnitus
* Metal implants in the head, neck or cochlea
* A pacemaker
* Migraines
* A history of taking medications that lower seizure threshold (i.e. such as tricyclic antidepressants or bupropion)
* Claustrophobia (due to the MRI)
* Used any form of tobacco in the past two years if they desire to be a non-smoking participant
* Plans to quit smoking in the next 30 days if they desire to be a smoking participant
* Current use of any medications for tobacco cessation (i.e. nicotine replacement, bupropion, varenicline, etc.)
* A report of a high motivation to quit smoking (score 7 or great on the Motivation scale)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Sheffer, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 11/4/2009 to 9/19/2011 from the surrounding community using primarily newspaper advertisements and word of mouth.
Pre-assignment Details: Enrolled participants were scheduled for an MRI of the head and needed to pass the MRI-screen (i.e., have no significant brain abnormalities) to continue with the study. Of the 49 participants who obtained an MRI, 6 participants did not pass this screen.
Groups:
- Smokers: Smokers were healthy adults between the ages of 19 and 55 years who had no intention of quitting smoking before the end of the study.
- Non-smokers: Healthy adult non-smokers who were between the ages of aged 19-55 years.
Period: Overall Study
Arm/Group | Smokers | Non-smokers
Started | 47 (75 passed telephone interview; 28 passed in-person interview, were enrolled, and sent for MRI.) | 19 (21 passed telephone interview; 19 passed the in-person interview, were enrolled, and sent for MRI.)
Completed | 16 (Completed three sessions of rTMS) | 14 (Completed three sessions of rTMS)
Not Completed | 31 | 5
Not completed — did not attend MRI | 14 | 3
Not completed — did not pass MRI screen | 6 | 0
Not completed — did not complete rTMS sessions | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smokers | Nonsmokers | Total
Number analyzed (Participants) | 47 | 19 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 19 | 66
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.38 (10.01) | 39.16 (11.21) | 41.45 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 33 | 7 | 40
Region of Enrollment [Number; unit: participants]
  United States | 47 | 19 | 66

OUTCOME MEASURES:

1. Primary Outcome: A Difference Score for the Log Value of K.
Description: K is a output value, a summary statistic, derived from a hyperbolic function that summarizes the rate at which monetary values are discounted according to the time they are received. The value of K can either increase or decrease from its baseline value. For example, an increase in K would indicate that the participant is choosing to receive larger amounts of money at a later point in time. A decrease would suggest the opposite - lesser amounts of money at an earlier point in time). The difference score is calculated from baseline to that immediately after 10 or 20 Hz rTMS.
Time Frame: baseline and immediately after stimulation, an average of 25 seconds.
Population: All participants that attended at least one session and provided at least some outcome data were included in the analyses
Measure: Log Mean (Standard Deviation); unit: log transformed values of K
Arm/Group | Smokers | Non-smokers
Number analyzed (Participants) | 23 | 16
log transformed values of K | -1.2215 (3.05) | -1.6742 (2.29)

ADVERSE EVENTS:
Arm/Group | Smokers | Non-smokers
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/19
Other Adverse Events (participants affected / at risk) | 0/47 | 0/19

LIMITATIONS AND CAVEATS:
We experienced significant subject attrition among smokers. We did not experience such attrition among nonsmokers. Also, six smokers were withdrawn because the MRI screen revealed brain abnormalities. No nonsmokers were withdrawn for this reason.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No